CLINICAL TRIAL: NCT05944666
Title: Standardization of the System of Multimodal Cognitive-motor Poststroke Rehabilitation, in Accordance With the Verification of Rehabilitation Potential, Rehabilitation Diagnosis and Patient Model, at the Stages of Medical Rehabilitation
Brief Title: Substantiation and Standardization of the Multimodal Cognitive-motor Rehabilitation System for Afterstroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine (Other)
Responsible Party: Principal Investigator, Nadezda Lyamina, Clinical Professor, Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3/15.05.2023
Record Dates: First submitted 2023-06-19; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Stroke Rehabilitation
Keywords: ischemic stroke rehabilitation; post-stroke dysfunction of the hand; cognitive disfunction; artificial intelligence; virtual reality; neurointerface; smart glove; biofeedback; cardiology risk control; lower limb medical rehabilitation; digital interactive technology; standartized rehabilitation technologies; verification of the rehabilitation potential

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Medical rehabilitation (MR) in acute period of IS-inpatient stage (Experimental): Devices Patients in acute period of IS receive a course of standart MR-program and in main group - rehabilitation with multimodal correction using and BFB-stabilometric training, cognitive-motor training in a virtual environment (VR), functional individually programmed stimulation of antagonist muscles of the lower limb (FES), subject-manipulative activity training to restore fine movements of the hand on a glove simulator, if moderate paresis of the upper limb - the neurointerface "Exokist-2" with EEG registration.
  Interventions: Procedure: Multimodal technology (MT); Procedure: Conventional rehabilitation
- MR in early recovery period of IS- inpatient stage (Experimental): Devices Patients in the early recovery period of IS receive a course of standart MR-program and in main group - rehabilitation with multimodal correction using and BFB-stabilometric training, cognitive-motor training in a virtual environment (VR), functional individually programmed stimulation of antagonist muscles of the lower limb (FES), subject-manipulative activity training to restore fine movements of the hand on a glove simulator, if moderate paresis of the upper limb - the neurointerface "Exokist-2" with EEG registration.
  Interventions: Procedure: Multimodal technology (MT); Procedure: Conventional rehabilitation
- MR in late recovery period of IS-inpatient stage (Experimental): Devices Patients in the late recovery period of IS receive a course of standart MR-program and in main group - rehabilitation with multimodal correction using and BFB-stabilometric training, cognitive-motor training in a virtual environment (VR), functional individually programmed stimulation of antagonist muscles of the lower limb (FES), subject-manipulative activity training to restore fine movements of the hand on a glove simulator, if moderate paresis of the upper limb - the neurointerface "Exokist-2" with EEG registration.
  Interventions: Procedure: Multimodal technology (MT); Procedure: Conventional rehabilitation
- MR in early recovery period of IS - outpatient stage (Experimental): Devices Patients in the early recovery period of IS receive a course of standart MR-program and in main group - rehabilitation with multimodal correction using and BFB-stabilometric training, cognitive-motor training in a virtual environment (VR), functional individually programmed stimulation of antagonist muscles of the lower limb (FES), subject-manipulative activity training to restore fine movements of the hand on a glove simulator, if moderate paresis of the upper limb - the neurointerface "Exokist-2" with EEG registration.
  Interventions: Procedure: Multimodal technology (MT); Procedure: Conventional rehabilitation
- MR in late recovery period of IS - outpatient stage (Experimental): Devices Patients in the late recovery period of IS receive a course of standart MR-program and in main group - rehabilitation with multimodal correction using and BFB-stabilometric training, cognitive-motor training in a virtual environment (VR), functional individually programmed stimulation of antagonist muscles of the lower limb (FES), subject-manipulative activity training to restore fine movements of the hand on a glove simulator, if moderate paresis of the upper limb - the neurointerface "Exokist-2" with EEG registration.
  Interventions: Procedure: Multimodal technology (MT); Procedure: Conventional rehabilitation

INTERVENTIONS:
Procedure: Multimodal technology (MT) — Only fo the patients of the Main group. It will be different programms depending on severety of UL or LL paresis. Patients will receive a course of rehabilitation with multimodal correction using BFB-stabilometric training, cognitive-motor training with double and triple tasks once a day for the affected hand, virtual reality, functional individually programmed stimulation of antagonist muscles of the lower limb (FES), subject-manipulative activity training to restore fine movements of the hand on a glove simulator, in moderate paresis of the upper limb, the neurointerface "Exokist-2" with EEG registration will be used. The program for IS patients includes 10 sessions in inpatient stage every day 15-30 min for the method, 15 sessions with the MT in outpatient stage: 15-30 minutes every method 2-3 times a week, 5-8 weeks.The total duration of one procedure is 2-3 hours.
Procedure: Conventional rehabilitation — It will be different programms depending on severety of UL or LL paresis. Conventional rehabilitation (CR) includes physiotherapy, kinesiotherapy, occupational therapy. The program for IS patients consists of 10 sessions of every day trainings for inpatients stage, 15 sessions with the CR for outpatient stage: 15-30 minutes every method 2-3 times a week, 5-8 weeks.The total duration of one procedure is 2-3 hours.

SUMMARY:
The aim of the study is to develop and scientifically substantiate a standardized system of multimodal cognitive-motor rehabilitation and its differentiated application in patients with cerebral stroke, according to verified rehabilitation potential based on the patient's rehabilitation model for the stages of medical rehabilitation, including inpatient-replacement technologies

DETAILED DESCRIPTION:
The object of the study The study will include 405 patients (men and women) with the diagnosis of ischemic stroke (IS) in the acute (0-21 day), early recovery (up to 6 months) and late recovery (6-12 months) periods with stato-locomotor disturbances, dysfunction (violation of neuromuscular movement control) of the upper limb (UL), lower limb (LL), mild or moderate cognitive impairment.

Patients will be randomly assigned to one of 6 experimental groups - 3 main groups of 70 patients each in the acute, early and late recovery period of IS and 3 comparison groups (each of 65 patients) in the acute, early and late recovery periods of IS. The patients in the main and comparison groups will be comparable in age, gender and symptoms.

Each participant of the study will be assigned an ordinal number. Patients of the main groups are planned to undergo a rehabilitation course with standardized multimodal correction, depending on the severity of functional and neuropsychological disturbances with the use of FBF-stabilometric training, cognitive-motor training with double and triple tasks in a virtual environment, functional individually programmed stimulation of antagonist muscles of the lower limb (FES), training of subject-manipulative activity for the restoration of fine hand movements on the glove simulator "SensoRehab"; when severe and moderate paresis of the upper limb, the neurointerface "Exokist-2" with EEG registration will be used.

The patients of comparison groups are planned to undergo a rehabilitation course with standart rehabilitation programms depending on the severity of functional and neuropsychological disturbances: kinesiotherapy, physical therapy, occupational therapy, massage.

The study is carried out at the inpatient stage, then patients are transferred to the outpatient stage of rehabilitation or controlled home self-rehabilitation using telemedicine technologies.

The mode of application of multimodal correction technology:

inpatient stage: 10 procedures every day (5 working days, 2 days the rest);the total duration of one procedure is 2-3 hours a day.

outpatient stage: 15 procedures, 2-3 times a week, the duration of the course is 5-8 weeks. The total duration of one procedure is 2-3 hours a day.

Multimodal correction technology will not be included in the rehabilitation program of patients in the comparison group.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 45 to 70 years after a first-onset IS, acute (1-21 days), early (22 days- 6 months), late recovery (6-12 months) periods.
* Supratentorial IS according to MRI of the brain.
* The severity of UL and LL paresis ranged from a score of 4 to 2 according to the Medical Research Council Scale (MRCS)
* Spasticity of 3 points or less by the Modified Ashworth Scale (MAS)
* Cognitive function more than 20 points on the Montreal Cognitive Assessment (MoCA)
* Affective disorders score less than 11 on the Hospital Anxiety and Depression Scale (HADS)
* The patient's ability and willingness to comply with the requirements of this protocol.

Exclusion Criteria:

1. Concomitant neurological diseases causing decreased muscle strength or increased muscle tone in the UL (e.g., cerebral palsy, brain injury).
2. Clinically significant limitation of the passive movement amplitude in the joints of the investigated hand, pronounced contracture and deformities of the upper extremity.
3. Use of other DIT, BFB techniques to restore impaired UL function within 30 days prior to the patient Inclusion Visit.
4. Severe visual impairment, decreased visual acuity of less than 0.2 in the worst eye according to the Golovin-Sivtsev Table24.
5. Sensory aphasia, gross motor aphasia.
6. Recurrent stroke.
7. Epilepsy
8. Unstable angina and/or heart attack in previous month.
9. Uncontrolled arterial hypertension.
10. Somatic diseases in decompensation stage.
11. Thrombosis of deep and superficial veins of the lower extremities
12. The presence of left-handedness in the patient according to the Edinburgh manual asymmetry questionnaire
13. Alcohol abuse, medical marijuana use or soft drug abuse within the 12 months prior to the Inclusion Visit.
14. Any medical condition, including mental disease or epilepsy that could affect the interpretation of study results, the study procedures or patient safety.

15 Pregnancy. 16. Lactation.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ICF motor and sensitive domains dynamic | Baseline, visit day 10 of inpatient rehabilitation, visit days 1, 7, 15 of MR in outpatient stage
  Changes in the severity of dysfunctions by at least 1 determinant point of at least 1 of the selected ICF domains characterizing motor stereotype, balance at rest and when walking, fine motor skills of the upper limb, sensory disorders, pain syndrome

SECONDARY OUTCOMES:
ICF cognitive and emotional domains dynamic | Baseline, visit day 10 of inpatient rehabilitation, visit days 1, 7, 15 of MR in outpatient stage
  Changes in the severity of disorders by at least 1 determinant point of at least 1 of the selected ICF domains characterizing neuropsychological disorders (cognitive, emotional) and personal factors.
Changes in level of impairment or dependence in daily life | Baseline, visit day 10 of inpatient rehabilitation, visit days 1, 7, 15 of MR in outpatient stage
  Changes of the degree of functional independence according to the Bartel index
Changes in Rankin scale | Baseline, visit day 10 of inpatient rehabilitation, visit days 1, 7, 15 of MR in outpatient stage
  Changes of the degree of disability, independence and rehabilitation outcomes according to the Rankin scale
Canges in Rehabilitation routing scale (RRS) | Baseline, visit day 10 of inpatient rehabilitation, visit days 1, 7, 15 of MR in outpatient stage
  Changes of the degree of disability, independence and rehabilitation outcomes according to the RRS
Changes of Life quality assessment | Baseline, visit day 10 of inpatient rehabilitation, visit days 1, 7, 15 of MR in outpatient stage
  Improving the quality of life according to the European Quality of Life Questionnaire EuroQol EQ-5D-5L
Changes of SF-36 questionnaire | Baseline, visit day 10 of inpatient rehabilitation, visit days 1, 7, 15 of MR in outpatient stage
  Changes of the quality of life scores according to the SF36

CONTACTS AND LOCATIONS:
Locations (1):
- Moscow Scientific and Practical Center of Medical Rehabilitation, Restorative and Sports Medicine, branch 3 and branch7, Moscow, Russia